CLINICAL TRIAL: NCT06993337
Title: Evaluation of Topical Bromelain Versus Topical Corticosteroids in Management of Recurrent Aphthous Stomatitis: A Randomized Controlled Trial
Brief Title: Effect of Topical Bromelain Versus Topical Corticosteroids in the Management of Recurrent Aphthous Stomatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Ayoub Mohamed, Master's Student in Oral Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMED 372
Record Dates: First submitted 2025-05-14; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Aphthous Stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Bromelains; Orabase; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 35% Topical Bromelain in Orabase (Experimental): Participants in this group will receive 35% bromelain gel incorporated into an orabase adhesive medium.
  Interventions: Dietary Supplement: 35% Topical Bromelain in Orabase
- 50% Topical Bromelain in Orabase (Experimental): Participants assigned to this group will be treated with 50% bromelain gel formulated in orabase.
  Interventions: Dietary Supplement: 50% Topical Bromelain in Orabase
- 0.1% Topical Triamcinolone Acetonide in Orabase (Active Comparator): This group will receive the standard treatment of 0.1% triamcinolone acetonide in orabase, commonly used for managing Recurrent Aphthous Stomatitis.
  Interventions: Drug: 0.1% Topical Triamcinolone Acetonide in Orabase

INTERVENTIONS:
Dietary Supplement: 35% Topical Bromelain in Orabase — Bromelain is a natural proteolytic enzyme derived from pineapple, recognized for its broad range of pharmacological properties. It exhibits significant anti-inflammatory effects by reducing edema. In addition to its anti-inflammatory activity, bromelain possesses antioxidant and analgesic properties.
  Arms: 35% Topical Bromelain in Orabase
Dietary Supplement: 50% Topical Bromelain in Orabase — Bromelain is a natural proteolytic enzyme derived from pineapple, recognized for its broad range of pharmacological properties. It exhibits significant anti-inflammatory effects by reducing edema. In addition to its anti-inflammatory activity, bromelain possesses antioxidant and analgesic properties.
  Arms: 50% Topical Bromelain in Orabase
Drug: 0.1% Topical Triamcinolone Acetonide in Orabase — Triamcinolone acetonide in orabase, a corticosteroid-based standard treatment for Recurrent Aphthous Stomatitis (RAS), is used for its strong anti-inflammatory and immunosuppressive effects. In this study, it serves as the conventional treatment against the novel therapy
  Arms: 0.1% Topical Triamcinolone Acetonide in Orabase

SUMMARY:
Bromelain, a natural product, exhibits anti-inflammatory, immunomodulatory, and wound-healing properties. However, its efficacy in treating oral mucosal ulcers remains unexplored. This study aims to evaluate the effect of bromelain as a safe alternate for management of RAS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Diagnosed with RAS.
* Onset of ulcer within the last 48 hours.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* History of hematological deficiencies, GIT disorders, Behcet's disease and major systemic diseases.
* Pregnant or breastfeeding patients.
* Previous treatment for the current ulcer episode.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain associated with ulcers | Recorded at baseline, day 2, day 4 and day 7
  Pain reduction will be measured using a visual analog scale (VAS). VAS is a self-reported pain scores ranging from 0 to 10

SECONDARY OUTCOMES:
Reduction in ulcer size | Recorded at baseline, day 2, day 4 and day 7
  The reduction in ulcer size will be assessed using periodontal probe to measure dimensions in millimeters (mm)
Number of oral ulcers | Recorded at baseline, day 2, day 4 and day 7
Healing time of oral ulcer | Recorded at baseline, day 2, day 4 and day 7
  The time to complete healing will be determined by the number of days until the ulcer is no longer visible upon clinical examination
Oral ulcer activity index | Recorded at baseline, day 2, day 4 and day 7
  Oral ulcer activity index will be measured by Composite index (CI). CI score (0-10) is calculated by summing of subscale scores of oral ulcer activity (0 vs 1), oral ulcer-related pain status evaluated by categorized VAS (0-5) and the mean global functional disability score evaluated by 5-point Likert-type scale (0-4)